CLINICAL TRIAL: NCT01957826
Title: Phase I/II Randomized Clinical Trial to Assess the Safety and Feasibility of Transendocardial Injection of Bone Marrow Autologous Mesenchymal Stem Cells in Patients With Idiopathic Dilated Cardiomyopathy.
Brief Title: Mesenchymal Stem Cells for Idiopathic Dilated Cardiomyopathy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Collaborators: Ministerio de Sanidad, Servicios Sociales e Igualdad (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FIBHGM-ECNC017-2010; 2010-024406-35 (EudraCT Number); MIYOCYTE (Other: MYOCYTE)
Record Dates: First submitted 2012-12-21; First posted 2013-10-08 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Primary Idiopathic Dilated Cardiomyopathy
Keywords: mesenchymal; stem cells; transendocardial injection; dilated idiopathic cardiomyopathy; idiopathic cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- placebo comparator (Placebo Comparator): transendocardial injection of placebo solution
  Interventions: Other: placebo intervention
- bone marrow-derived MSCs injection (Experimental): transendocardial injection of 30-40 million bone marrow-derived MSCs with the NOGA XPTM platform. 15 injections in the anterior wall of the left ventricle.
  Interventions: Other: bone marrow-derived MSCs injection

INTERVENTIONS:
Other: bone marrow-derived MSCs injection — transendocardial injection of 30-40 million bone marrow-derived MSCs with the NOGA XPTM platform. 15 injections in the anterior wall of the left ventricle.
  Arms: bone marrow-derived MSCs injection
Other: placebo intervention — placebo administration
  Arms: placebo comparator

SUMMARY:
The purpose of this study is to assess the safety, the feasibility and the efficacy of transendocardial injection of bone marrow-derived mesenchymal stem cells (MSCs) in patients with dilated idiopathic cardiomyopathy.

DETAILED DESCRIPTION:
Chronic congestive heart failure (CHF) is a public health problem that entails high rates of morbidity and mortality, and enormous costs for health systems worldwide. In the United States there are 5 million people living with CHF, and each year 60.000 people reach terminal phases of the disease, with mortality rates of 70-80% at two years. Although the first cause of CHF in developed countries is atherosclerotic coronary artery disease (CAD), dilated idiopathic cardiomyopathy (DCM) represents almost half of the cases of newly diagnosed CHF. Treatment of CHF includes pharmacological and non-pharmacological strategies, including implantable cardioverter defibrillators, cardiac resynchronization therapy and heart transplantation. Despite all these advances, CHF prognosis remains poor. Cardiac stem cell therapy emerged more than ten years ago as a new hope for CHF patients.

Although the most extensive evidence of the benefits of stem cell therapy for cardiovascular diseases refers to ischemic heart disease (CAD), initial experiences with stem cells for other conditions such as DCM are encouraging.

This randomized clinical trial will include 70 patients with DCM, left ventricular ejection fraction (LVEF) between 20% and 45%, and who are symptomatic in New York Heart Association (NYHA) functional class II-III/IV. In a first-in-man pilot phase, 10 patients will be treated with transendocardial injections of bone marrow-derived MSCs after cardiac catheterization and NOGA XPTM mapping of the left ventricle. A Data and Safety Monitoring Board (DSMB) will analyse the safety and feasibility of this first phase of the trial, and then 60 patients more will be randomized to receive MSCs or placebo (ratio 3:1).

Primary objectives include safety and feasibility variables, and secondary objectives include efficacy variables. All patients will be studied with a complete cardiac imaging protocol that includes: electrocardiography, echocardiography, treadmill tests with oxygen consumption, holter, laboratory analyses, magnetic resonance imaging (MRI), single photon emission computed tomography (SPECT), electromechanical mapping (NOGA XPTM) and quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* II-III NYHA functional class, under optimal medical therapy.
* LVEF ≥ 20% and ≤ 45% by echocardiography, SPECT or left ventriculogram one month prior to enrollment.
* Anterior wall thickness ≥ 8 mm by echocardiography or MRI one month prior to enrollment.
* Idiopathic DCM diagnosis (having excluded CAD, valvular heart disease, cardiac toxic drugs, tachyarrhythmias, metabolic diseases, systemic diseases, infectious diseases) six months prior to enrollment.
* Patients rejected for heart transplantation should have been discussed in the Heart Team at their respective centres, and a document stating the reason for exclusion will be kept in the medical record.
* Able to exercise on a treadmill, MVO2 between ≥ 12 and ≤ 21 ml/Kg/min.
* Hemodynamic stability (blood pressure > 100/40 mmHg, heart rate < 110 bpm and oxygen saturation > 95%).
* Negative pregnancy test in women.
* Signed informed consent

Exclusion Criteria:

* Evidence of secondary dilated cardiomyopathy causes: CAD, valvular heart disease, cardiac toxic drugs, tachyarrhythmias, metabolic diseases, systemic diseases, infectious diseases, myocarditis or postpartum ventricular dysfunction.
* Permanent atrial fibrillation.
* Candidates for ICD or CRT devices. Patients with theses devices can be enrolled if the device has been implanted at least 6 months before inclusion, and only if no-response has been observed to CRT.
* Candidates for heart transplantation if surgery is anticipated in the next 2 years.
* Left ventricular thrombus by echocardiography, MRI or left ventriculogram.
* Peripheral artery disease that precludes cardiac catheterization with 8 Fr sheaths. .
* Anterior wall thickness < 8 mm by echocardiography or MRI one month prior to enrollment.
* Chronic renal failure (creatinine > 2,5 mg/dL).
* I or IV NYHA functional class. Cardiogenic shock is defined as systolic blood pressure < 90 mmHg with no response to fluids, or < 100 mmHg with inotropes and without bradycardia.
* Previous history of drug abuse (alcohol, etc…).
* Acute or chronic infectious disease (including B/C hepatitis and HIV).
* Pregnancy or child-bearing period.
* MRI contraindications: pacemakers, ICD, metalic prosthesis, etc.
* Bleeding or coagulation disorders (INR > 2 without anticoagulation treatment).
* Cancer history 5 years prior to enrollment.
* Life expectancy less than 1 year.
* Any disease or condition that the investigator finds decisive for exclusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2013-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac adverse events. SAEs and AEs. | change from enrollment( 1, 3, 6, 12, 18 and 24 months)
  Major adverse cardiac adverse events includes cerebral adverse events
NYHA functional class. | Change from enrolment( 1, 3, 6, 12, 18, 24 months)
Incidence of complications with the use of NOGA XPTM catheters. | Change from enrolment( 1, 3, 6, 12, 18, 24 months)
Laboratory parameters including C-reactive protein an brain natriuretic peptide | Change from enrolment( 1, 3, 6, 12, 18, 24 months)

SECONDARY OUTCOMES:
NYHA Functional Class | 1, 3, 6, 12, 18, 24 months
Max.oxygen consumption(MVO2),functional capacity. | 6,12,24 months
Quality of life questionnaires | 6,12 and 24 months
  include 36-item Short Form Survey(SF 36) and Minnesota Living UIT Heart Failure questionnaire
Extension. of perfusion defects(MRI/SPECT). | 6 and 24 months
LVEF, ventricular vol.,wall motion score index(echocard./MRI/SPECT | 6,12 and 24 months
LVEF(left ventriculogram, electromech. mapping parameters(NOGA XPTM)) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Fernandez Aviles, PhD, Study Chair — Hospital General Universitario Gregorio Marañón
Locations (2):
- Spain (2):
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Clinico Universitario de Valladolid, Valladolid, Valladolid